CLINICAL TRIAL: NCT02916979
Title: A Pilot Trial Examining Myeloid-Derived Suppressor Cells and Checkpoint Immune Regulators' Expression in Allogeneic Stem Cell Transplant Recipients Using Myeloablative Busulfan and Fludarabine
Brief Title: Myeloid-Derived Suppressor Cells and Checkpoint Immune Regulators' Expression in Allogeneic SCT Using FluBuATG
Acronym: FluBuATG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Kenneth Meehan, Director, Bone Marrow Transplant Program, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D16127
Record Dates: First submitted 2016-08-15; First posted 2016-09-28 (Estimated); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Leukemia, Lymphoid; Leukemia, Myeloid; Myelodysplastic Syndromes; Myelofibrosis; Lymphoma, Malignant; Multiple Myeloma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Leukemia, Lymphoid; Leukemia, Myeloid; Myelodysplastic Syndromes; Primary Myelofibrosis; Lymphoma; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — fludarabine; Busulfan; thymoglobulin; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Conditioning Regimen (Other): Fludarabine, Busulfan, Rabbit ATG, Methotrexate
  Interventions: Drug: Fludarabine; Drug: Busulfan; Biological: Rabbit ATG; Drug: Methotrexate

INTERVENTIONS:
Drug: Fludarabine — Fludarabine: 30 mg/m2 daily for 5 days
Drug: Busulfan — Busulfan: 100 mg/m2 daily for 4 days
Biological: Rabbit ATG — Rabbit ATG:
  Related donors: 1.5 mg/kg daily x 2 days (on days -6 and -5) Unrelated donors: 1.5 mg/kg on day - 6 2 mg/kg on day -5 2.5 mg/kg on day -4
Drug: Methotrexate — Methotrexate:
  Related donors: 5 mg/m2 on days 1, 3 and 6 Unrelated donors: 5 mg/m2 on days 1, 3, 6 and 11

SUMMARY:
This study is examining a chemotherapy regimen and immune suppressive medications in the setting of an allogeneic stem cell transplant. A pilot clinical trial to characterize the incidence, prevalence and function of myeloid-derived suppressor cells (MDSCs) and immune checkpoint regulators (V-domain Ig Suppressor of T-cell Activation [VISTA], cytotoxic T-lymphocyte- associated protein 4 [CTLA-4], programmed death-ligand 1 [PD-L1]) during early immune recovery following an allogeneic stem cell transplant. The site will use a myeloablative regimen of fludarabine with busulfan, adopted from CALGB 100801, to define clinical endpoints, including engraftment, 100 day survival and one year survival (Objective #1). The site will characterize the incidence, prevalence and function of MDSCs and immune checkpoint regulators in patients' blood and bone marrow following transplantation (Objective #2). The site will correlate these laboratory results with clinical outcomes and the incidence of graft-versus-host disease (GVHD). As an exploratory aim, in those patients experiencing GVHD and requiring treatment, the site will define the MDSCs frequency and checkpoint regulator expression and correlate these results with the patient's response to GVHD therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age less than or equal to 75 years
2. The patient must be approved for transplant by the treating transplant physician. This includes completion of their pretransplant workup, as directed by standard Dartmouth-Hitchcock Medical Center (DHMC) Standard Operating Procedures (SOPs). DHMC SOP for Pretransplant Evaluation of allogeneic recipient.
3. The patient must have a disease, listed below, with treatment responsiveness that the treating transplant physician believes will benefit from an allogeneic stem cell transplant. The diseases include:

   1. Acute leukemia AML (Acute Myeloid Leukemia), ALL (Acute Lymphoid Leukemia)
   2. Chronic leukemia CML (Chronic Myeloid Leukemia), CLL (Chronic Lymphoid Leukemia)
   3. Myelodysplasia
   4. Myelofibrosis
   5. Lymphoma NHL (Non-Hodgkin's Lymphoma) and Hodgkin's disease
   6. Plasma cell disorder, including myeloma, Waldenstrom's Macroglobulinemia
4. Donor availability- the patient must have an identified donor

   1. Sibling Availability of a 6 out of 6 identical donor
   2. Unrelated donor: Availability of a 6 out of 6 unrelated donor
5. No human immunodeficiency virus (HIV) infection or active hepatitis B or C
6. Easter Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
7. Diffusing capacity of the lungs for carbon monoxide DLCO more than or equal to 40 percent predicted
8. Left ventricular ejection fraction more than or equal to 35 percent
9. Serum bilirubin less than 2x upper limit of normal transaminases less than 3x normal at the time of transplant
10. No active or uncontrollable infection
11. In female, a negative pregnancy test if experiencing menstrual periods
12. No major organ dysfunction precluding transplantation
13. No evidence of an active malignancy that would limit the patient's survival to less than 2 years. If there is any question, the principal investigator can make a decision.

Exclusion Criteria:

1. Psychiatric disorder or a mental deficiency of the patient that is sufficiently severe to make compliance with the treatment unlikely, and making informed consent impossible.
2. Major anticipated illness or organ failure incompatible with survival from bone marrow transplant.
3. History of refractory systemic infection

Donor eligibility

1. Human leukocyte antigen (HLA) 6 out of 6 matched related or unrelated donor.
2. The donor must be healthy and must be willing to serve as a donor, based on standard guidelines
3. The donor must have no significant comorbidities that would put the donor at marked increased risk
4. There is no age restriction for the donor
5. Informed consent must be signed by donor, if sibling donor, or by third party if unrelated donor.

   Donor Exclusion Criteria
6. The National Marrow Donor Program (NMDP) guidelines for exclusion criteria will be used. In addition, the following donors are NOT eligible:
7. Syngeneic donor
8. Pregnant or lactating donor
9. Human immunodeficiency virus (HIV) or active HepB or C in the donor
10. Donor unfit to receive Granulocyte-colony stimulating factor (GCSF) and undergo apheresis
11. A donor with a psychiatric disorder or mental deficiency that makes compliance with the procedure unlikely and informed consent impossible

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09-06 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Number of patients who are surviving at 100-Days post-transplant | 100 Days
  100-Day survival of patients

SECONDARY OUTCOMES:
Time to marrow engraftment | 100 Days
  Time to marrow engraftment (defined as absolute neutrophil count > 500/mm3 and platelets > 20,000/mcl for three consecutive days (count first day as engraftment)
Assessing all subjects' response to treatment at 100 days post-transplant | 100 Days
  Response to treatment at 100 days using standard international response criteria, based on CIBMTR definitions.
Assessing all subjects' response to treatment at 1 year post-transplant | 365 Days
  Response to treatment at one year using standard international response criteria, based on CIBMTR definitions.
Assessing all subjects' survival at 1 year post-transplant | 365 Days
  One year survival
Assessing the mortality rate of patients in the first 100 days post-transplant | 100 Days
  Treatment-related mortality in the first 100 days
Assessing the number of treatment-related adverse events | 365 Days
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Collecting the incidents of GvHD experienced by patients post-transplant | 365 Days
  Incidence of acute and chronic GVHD
Assessing the donor-chimerism at 30, 60 and 90 days post-transplant | 30, 60, and 90 Days
  Donor-recipient chimerism following transplant at Days 30, 60 and 90.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Meehan, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No